CLINICAL TRIAL: NCT04387292
Title: Ocular Sequelae of Patients Hospitalized for Respiratory Failure During the COVID-19 Epidemic
Acronym: SOCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MMT_2020_12
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2021-08

CONDITIONS: COVID19; Ophthalmopathy
Keywords: COVID19
MeSH Terms: conditions — COVID-19; Eye Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ophthalmologic exam (Experimental)
  Interventions: Procedure: Ophthalmologic exam

INTERVENTIONS:
Procedure: Ophthalmologic exam — * Visual acuity (ETDRS exam)
  * Slit lamp examination : fluorescein test, Oxford score, break up time, Schirmer II test
  * Lipiview
  * Eye pressure measurement (air tonometer)
  * Wide field retinophotography
  * Multicolor and auto-fluorescence retinophotography
  * Indocyanine green retinal angiography
  * Optical coherence tomography (OCT) B posterior pole scan
  * OCT Angiography (OCT-A) of the optic nerve and posterior pole
  * Adaptive optics
  * Visual field (Humphrey)

SUMMARY:
Ophthalmologic damages secondary to COVID-19 coronavirus infection are little described. The ocular involvement is probably multiple, ranging from pathologies of the anterior segment such as conjunctivitis and anterior uveitis to disorders that threaten vision such as retinitis or optic neuropathy. On the other hand, in addition to this impairment, when patients are hospitalized for acute respiratory failure, complications related to possible resuscitation, medication prescriptions, positioning and oxygenation.

COVID-19 itself, has several components:

* An apoptotic action of the viral attack which will generate cellular destruction, whether pulmonary, cardiac or renal or maybe ocular
* A secondary autoimmune action with the development of major vascular inflammation, possibly reaching the retinal, choroidal, and optic nerve vessels. A secondary "hyper" inflammatory syndrome with flashing hypercytokinemia and multi-organ decompensation is described in 3,7% to 4 ,3% of severe cases.
* A thromboembolic action

DETAILED DESCRIPTION:
Upon discharge from hospital for COVID-19 infection (or during a telephone call for patients already discharged at the start of the study), patients will be informed of the study. An ophthalmology appointment will be given to them between 4 and 6 months after their discharge.

During the ophthalmology appointment, the patient's clinical data will be collected during an interview (medical and treatment history, blood group). The patient will benefit from a full ophthalmological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients having been hospitalized for a confirmed COVID-19 infection (CT-scanner or PCR- Polymerase chain reaction)

Exclusion Criteria:

* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Description of the ophthalmological problems observed | 6 months after discharge of hospitalization
  Multimodal ophthalmologic imaging

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France, France

REFERENCES:
- [Result] Abdelmassih Y, Azar G, Bonnin S, Scemama Timsit C, Vasseur V, Spaide RF, Behar-Cohen F, Mauget-Faysse M. COVID-19 Associated Choroidopathy. J Clin Med. 2021 Oct 13;10(20):4686. doi: 10.3390/jcm10204686. PMID 34682810